CLINICAL TRIAL: NCT02193685
Title: Identification of Genetic, Immunologic and Microbial Markers of Hirschsprung Associated Enterocolitis in Children With Hirschsprung Disease
Brief Title: Identification Genetic, Immunologic and Microbial Markers of Hirschsprung Associated Enterocolitis in Children With Hirschsprung Disease
Acronym: HAEC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Karolinska University Hospital (Other); Children's Hospital Los Angeles (Other); UCSF Benioff Children's Hospital Oakland (Other); University of Michigan (Other); The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Philip K. Frykman, MD, PhD, MBA, Associate Director, Pediatric Surgery, Cedars-Sinai Medical Center
Other Study IDs: Biomarkers of HAEC
Record Dates: First submitted 2014-07-09; First posted 2014-07-18 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-08

CONDITIONS: Hirschsprung Disease; Enterocolitis
Keywords: (HAEC) Hirschsprung Associated Entrocolistis; (HD) Hirschsprung Disease; (IBD) Inflammatory Bowel Disease; Children
MeSH Terms: conditions — Hirschsprung Disease; Enterocolitis; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Procedures include prospective data collection from medical records venipuncture and stool collection. 4 cc of blood will be drawn at the screening visit for genetic and immune testing. Additional 8.5 cc of blood will be drawn for CSMC patients for establishment of cell lines.
  1. Stool sample collected at screening or follow-up if patient unable to provide at screening.
  DNA will be prepared from blood for Genome Wide Association Study and mutational analysis 2. Serological immune markers for inflammatory bowel disease (IBD) including ANCA, ASCA, OMPC, I2, and CBir1 and any newly identified markers. These tests will only be performed on patients who consent to the immune response sub-study. No additional blood sample required. 3. Collect and store fresh fecal specimens for future evaluation by molecular methodologies to determine relative proportions of enteric microflora.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Subjects with HAEC: There is no intervention involvement. The clinical data and biologic specimens collected during the study will serve as an invaluable resource for a wide spectrum of clinical and translational ancillary studies directly related to the aims and goals of the study.
- Subjects without HAEC: A subgroup of children who have Hirschsprung Disease may or may not develop enterocolitis; therefore we will be identifying the bio-markers in children with or without associated enterocolitis.

SUMMARY:
To identify demographic, clinical, genetic, immunologic and/or microbial (i.e., fecal stream characterization) risk factors that influence the likelihood of development of the HAEC phenotype in children who carry the diagnosis of HD. The newly formed HAEC Collaborative Research Group (HCRG) will utilize the 4 participating centers in the current consortia and recruit additional centers to enroll children diagnosed with Hirschsprung disease.

1a: To recruit 200 patients with Hirschsprung disease without HAEC.

1b: To recruit 200 patients with Hirschsprung disease and HAEC using standardized diagnostic criteria by collaborating with participating members of the HAEC Collaborative Research Group[1].

1c: To collect clinical and demographic information from well-characterized HD patients both with and without HAEC.

1d: To collect samples blood for DNA for genome wide association study (GWAS) by high throughput SNP technology and mutational analysis of known HSCR genes.

1e: To collect serum samples at the time of recruitment in a subset cohort (n=50 HD only, n=50 HD + HAEC) for serological immune markers known for inflammatory bowel disease (IBD) including ANCA, ASCA, OMPC, I2, and CBir1 and any newly identified markers.

1f: To collect and store fresh fecal specimens for future evaluation by molecular methodologies to determine relative proportions of enteric microflora in a subset cohort (n=50 HD only, n=50 HD + HAEC) of children (<18 years).

1g: To establish a Centralized Data Coordinating Center for data collection, data quality and detailed data analyses (CSMC) and tissue bank (CSMC) to facilitate specimen analysis for this study.

The HAEC risk factor identification will be completed by multivariate logistic regression analysis. Genetic association will be studied for each SNP in the GWAS together with all other potential risk factors. Further analysis will be carried out to evaluate multiple SNPs/genes simultaneously.

DETAILED DESCRIPTION:
Emerging data suggests that the distinct phenotype of HAEC in children with HD may be the result of the complex interplay between host genetics, immune response and environmental triggers. Data suggest that approximately 20-30 percent of patients with HD develop HAEC. Thus, well-designed, multi-disciplinary investigations of genetic, immune and microbial etiologies of HAEC, with sufficient power to detect differences in disease phenotype are critically needed.

The Hirschsprung Disease clinical phenotype of HAEC:

Hirschsprung disease (HD; also known as congenital aganglionic megacolon) affects 1 in 5000 live births [2]. Surgical repair (excision of the aganglionic colon and pull through of the normally ganglionated intestine to the anal canal) is typically performed in infants with HD during the first few months of life [3, 4]. A subgroup of these children with HD will also develop Hirschsprung associated enterocolitis (HAEC), a potentially severe infection of the small bowel and colon[5]. Children who develop HAEC can present with fever, abdominal distention, explosive diarrhea, vomiting, lethargy, and if not diagnosed and treated promptly, can lead to life threatening sepsis and death. HAEC may occur pre- or post-surgery in HD patients. There have been widely varying reports of HAEC incidence ranging from 15-50% pre-surgery to 2-30% post-surgery. A lack of clear definition of HAEC criteria is at least partially responsible for this significant variation in reported incidence[6, 7]. A standardized definition of HAEC was recently developed and published in 2009[1]. The HAEC score consists of the most important clinical diagnostic criteria for HAEC identified from a group of international experts using the Delphi method. Preliminary validation with case scenarios was achieved and the HAEC score can now be used as a standardized and reproducible outcome measure for future studies on children with Hirschsprung disease. Now it is possible to perform rigorous studies of the genetic, immune, and microbial differences in HD patients who develop HAEC compared with those children with HD that have not developed HAEC.

Genetic variation: Currently there are 10 different genes identified (RET, GDNF, NTN, EDNRB, ET3, ECE-1, SOX10, ZFHX1B, PHOX2B, NGR1) in individuals affected with either isolated or syndromic Hirschsprung disease. The RET gene plays a critical role in ENS development and mutations in the RET gene have been found in 7-35% of sporadic cases and approximately 50% of familial cases. EDNRB and ET3 each account for approximately 5% of patients with HD and also are responsible for Shah-Waardenberg Syndrome. Mutations in each of the remaining 7 genes have been found in a small number of isolated and syndromic HD patients[8].

The RET tyrosine kinase signaling pathway plays a major role in ENS migration, along with its ligands GDNF and NTN. The EDNRB G-protein coupled receptor together with its ligand ET3 and endothelin cleavage enzyme ECE-1 forms a separate signaling pathway important in ENS development. The RET and EDNRB signaling pathways appear interact with an additive effect through an as yet to be described mechanism. PHOX2B is a transcriptional regulator of the RET gene and SOX10 appears to be a transcriptional regulator of both RET and EDNRB genes. The complex regulation of the genes in each pathway, combined with the cross-signaling between pathways and the effects on ENS migration is the subject of ongoing investigations[8, 9].

Current thought is that while some HD patients have a single mutation that is sufficient to cause HD, many patients likely have weaker mutations in multiple HD susceptibility genes that together are sufficient to cause HD[8, 9]. While there has been intense study of the genetics of HD over many years, there has been no attention given to possible genetic etiologies of HAEC. To date, the influence of genotype on the HAEC phenotype has received little attention, thereby providing additional merit for this proposal.

Immune markers and HAEC phenotypes:

One hypothesis is that HAEC may result from differing immune responses to microbial antigens in HD patients as has been found in patients with inflammatory bowel disease. Antibodies to the E. coli outer-membrane porin C (OmpC), the Pseudomonas fluorescens CD related protein (I2), anti CBiR1 (anti-flagellin), as well as Saccaromyces cerevisiae (ASCA) and autoantigens, perinuclear anti-neutrophil antibody (pANCA) are known to be elevated in the patients diagnosed with Crohn Disease (CD) and ulcerative colitis (UC). Established patterns of elevation of these antibodies serve as very important tools in establishing a diagnosis of IBD, as well as distinguishing patients with UC from those with CD.

By contrast, HAEC is a relatively poorly studied intestinal inflammatory disorder in children with clinical features similar to pediatric IBD. At present little attention has been given to the exploring the similarities in immune responses in HAEC patients to IBD patients. Our aim is to measure a panel of antibodies routinely used for IBD patients, and compare HD patients with and without HAEC. One or more antibody levels may serve as a biomarker for HD patients at risk of developing HAEC.

Microbial factors:

Data suggest that altered gut microbial populations may be partially responsible for the development of HAEC in susceptible HD patients. Most studies have focused on Clostridium difficile, because two groups reported increased frequency of C. diff. toxin positive stools in HD patients with HAEC compared with those without HAEC .[10, 11] Other groups subsequently reported very low frequencies of C. diff. toxin positivity in their patients with HAEC, thereby calling into question the role C. diff. plays in the pathogenesis of HAEC.[12] Other investigators have found E. coli, C. diff. and Cryptosporidium adherent to enterocytes on histological examinations of colon biopsies of patients with HAEC.[5] These findings indicate a breech in the protective mucus gel layer covering the luminal surface of the colon, leading to invasion of the epithelial barrier. Taken together, these studies suggest that the intestine-microbial interaction may be important in the pathogenesis of HAEC.

Moreover, the study of intestine-microbial interactions which lead to development of HAEC might best be undertaken in the pediatric patient whereby influences of host fecal microbial constituents are more easily elucidated. Therefore, research must not fail to identify other critically important pathogens by too narrow a focus on only known pathogens residing in colonic fecal streams in the genetically susceptible host. In addition, the characterization of gut microflora (i.e., fecal streams) and risk assessment of children with HD can optimally be done with a careful evaluation of both components - host and microbe in the index case. Successfully confirming or disproving infectious hypotheses requires that valid diagnostic tools be employed. Systematic investigations into potential infectious etiologies or normal enteric flora triggers of HAEC, therefore appear biologically plausible, and highly justified.

University of Michigan will be conducting metabolomics anaylsis of stool in children with Hirschsprung Disease. The analysis is focused on fatty acids metabolized by bacteria and yeast in the colon. The technique will use a GC-MASS SPEC approach to evaluate for pro-inflammatory vs. anti-inflammatory fatty acids in the stool of children with and or without Hirschsprung Associated Enterocolitis.

ELIGIBILITY:
Inclusion Criteria:

* 1. Males and females of all ages with a confirmed diagnosis of HD based on standardized histological criteria. Only Males and females ages 0 to 17 with a confirmed diagnosis of HD based on standardized histological criteria will be enrolled at CSMC.
* 2. Able to provide written informed assent if between the ages of 7 and 17. If age 6 and under, able to participate with parental permission.
* 3. Have consented to have specimens tested for genetics, immune responses, stool microflora.

Case Ascertainment:

All patients with a confirmed diagnosis of HD are eligible for enrollment. A diagnosis of HD for this study will require:

* 1)Documented histopathology showing absence of ganglion cells and is consistent with the diagnosis of HD.

Exclusion Criteria:

* 1. Intestinal neuronal dysplasia
* 2. Pseudo-obstruction

Ages: 1 Day to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with Hirschsprung disease under the age of 17 years.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2010-02; Primary Completion 2022-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
To identify genetic associations in HD patients who display HAEC phenotype | 7 years
  Rationale & hypothesis:
  Currently there is no generally accepted pathogenic hypothesis for Hirschsprung Associated Enterocolitis. A number of hypotheses propose the role of host genetics, host immune responses, and environmental factors such as microbial triggers, including in particular, enteric flora, resulting in disease susceptibility and development. These factors (host immune/inflammatory cells, intestinal epithelia and microbial flora) and their interactions may also be important determinants of disease phenotype and disease progression. Therefore we hypothesize that there are identifiable immunologic, genetic, enteric flora profiles along with clinical risk factors that influence development of HAEC phenotype.

SECONDARY OUTCOMES:
To identify immunological markers in HD patients who display HAEC phenotype | 8 years
  There is recent evidence that some HD patients who were thought to have refractory HAEC, actually developed IBD. Levin, DN et al. JPGN 2012. This aim is to explore the possibility that there may be similarities between the immune mechanisms involved in HAEC and IBD.

OTHER OUTCOMES:
To identify microbial markers in HD patients who display HAEC phenotype | 8-10 years
  Data suggest that altered gut microbial populations may be partially responsible for the development of HAEC in susceptible HD patients. Most studies have focused on Clostridium difficile, because two groups reported increased frequency of C. diff. toxin positive stools in HD patients with HAEC compared with those without HAEC .[10, 11] Other groups subsequently reported very low frequencies of C. diff. toxin positivity in their patients with HAEC, thereby calling into question the role C. diff. plays in the pathogenesis of HAEC.[12] Other investigators have found E. coli, C. diff. and Cryptosporidium adherent to enterocytes on histological examinations of colon biopsies of patients with HAEC.[5] These findings indicate a breech in the protective mucus gel layer covering the luminal surface of the colon, leading to invasion of the epithelial barrier. Taken together, these studies suggest that the intestine-microbial interaction may be important in the pathogenesis of HAEC.

CONTACTS AND LOCATIONS:
Overall Officials: Philip K Frykman, MD, PhD, MBA, Principal Investigator — Associate Professor, Surgery and Biomedical Sciences Associate Director, Pediactic Surgery for Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center 8723 Alden Drive, Suite 240, Los Angeles, California, United States

REFERENCES:
- [Background] Frykman PK, Cheng Z, Wang X, Dhall D. Enterocolitis causes profound lymphoid depletion in endothelin receptor B- and endothelin 3-null mouse models of Hirschsprung-associated enterocolitis. Eur J Immunol. 2015 Mar;45(3):807-17. doi: 10.1002/eji.201444737. Epub 2015 Jan 19. PMID 25487064
- [Background] Frykman PK, Short SS. Hirschsprung-associated enterocolitis: prevention and therapy. Semin Pediatr Surg. 2012 Nov;21(4):328-35. doi: 10.1053/j.sempedsurg.2012.07.007. PMID 22985838
- [Result] Demehri FR, Frykman PK, Cheng Z, Ruan C, Wester T, Nordenskjold A, Kawaguchi A, Hui TT, Granstrom AL, Funari V, Teitelbaum DH; HAEC Collaborative Research Group. Altered fecal short chain fatty acid composition in children with a history of Hirschsprung-associated enterocolitis. J Pediatr Surg. 2016 Jan;51(1):81-6. doi: 10.1016/j.jpedsurg.2015.10.012. Epub 2015 Oct 22. PMID 26561246
- [Result] Frykman PK, Nordenskjold A, Kawaguchi A, Hui TT, Granstrom AL, Cheng Z, Tang J, Underhill DM, Iliev I, Funari VA, Wester T; HAEC Collaborative Research Group (HCRG). Characterization of Bacterial and Fungal Microbiome in Children with Hirschsprung Disease with and without a History of Enterocolitis: A Multicenter Study. PLoS One. 2015 Apr 24;10(4):e0124172. doi: 10.1371/journal.pone.0124172. eCollection 2015. PMID 25909773
- [Derived] Frykman PK, Patel DC, Kim S, Cheng Z, Wester T, Nordenskjold A, Kawaguchi A, Hui TT, Ehrlich PF, Granstrom AL, Benliyan F; HAEC Collaborative Research Group (HCRG). Inflammatory Bowel Disease Serological Immune Markers Anti-Saccharomyces cerevisiae Mannan Antibodies and Outer Membrane Porin C are Potential Biomarkers for Hirschsprung-associated Enterocolitis. J Pediatr Gastroenterol Nutr. 2019 Aug;69(2):176-181. doi: 10.1097/MPG.0000000000002358. PMID 30964819